CLINICAL TRIAL: NCT01121406
Title: Phase II Randomized Trial of the Polo-like Kinase 1 Inhibitor BI 6727 Monotherapy Versus Investigator´s Choice Chemotherapy in Ovarian Cancer Patients Resistant or Refractory to Platinum-based Cytotoxic Therapy
Brief Title: BI 6727 (Volasertib) Randomised Trial in Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1230.18; 2009-015770-35 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-04-13; First posted 2010-05-12 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-07

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Gemcitabine; Topotecan; liposomal doxorubicin; BI 6727

ARMS (2):
- BI 6727 (Experimental): Patients receive BI 6727 infusion every 3 weeks
  Interventions: Drug: BI 6727
- Cytotoxic (Active Comparator): At the investigator discretion, patient will receive one of the following cytotoxics: topotecan, paclitaxel, gemcitabine or liposomal doxorubicin
  Interventions: Drug: Paclitaxel; Drug: Gemcitabine; Drug: Topotecan; Drug: Pegylated liposomal doxorubicin (PLD)

INTERVENTIONS:
Drug: Paclitaxel — Patients receive paclitaxel in a 4 week schedule
  Arms: Cytotoxic
Drug: Gemcitabine — Patients receive gemcitabine in a 3 week schedule
  Arms: Cytotoxic
Drug: Topotecan — Patients receive topotecan in 3 or 4 week schedule
  Arms: Cytotoxic
Drug: Pegylated liposomal doxorubicin (PLD) — Patients receive PLD in a 4 week schedule
  Arms: Cytotoxic
Drug: BI 6727 — Patients receive BI 6727 infusion every 3 weeks
  Arms: BI 6727

SUMMARY:
This is an international, randomized phase II trial. The aim is to assess the efficacy and the safety of BI 6727 Versus investigator's best choice single agent cytotoxic in recurrent third and fourth lines platinum resistant/refractory ovarian cancer.

100 patients will be randomised at the study entry to receive either BI 6727 (Arm A: 50 patients) or non-platinum single agent cytotoxic (Arm B: 50 patients) Treatment will be continued until disease progression or unacceptable toxicity. Primary endpoint: disease control rate at week 24 according to Response Evaluation Criteria In Solid Tumours version 1.1.

Secondary endpoints: efficacy (progression free survival, overall survival, biological tumour response, biological progression free survival assessed by serum CA 125 according to Gynecologic Cancer Intergroup criteria, safety according to the NCI CTCAE v.3, disease symptoms control assessed by the EORTC QLQ-C30, QLQ-OV28 and individual symptoms questionnaires, pharmacokinetics of BI 6727.

Others endpoints: biomarkers and pharmacogenetics analysis (optional)

ELIGIBILITY:
Inclusion criteria:

1. Confirmed recurrent epithelial ovarian carcinoma, peritoneal carcinoma or fallopian tube carcinoma.
2. Platinum resistant or platinum refractory disease.
3. Eastern Collaborative Oncology Group performance status < = 2.
4. Life expectancy > = 3 months.
5. At least one measurable lesion (Response Evaluation Criteria In Solid Tumours version 1.1).
6. Adequate hepatic, renal and bone marrow functions.
7. signed written informed consent prior to admission to the study.

Exclusion criteria:

1. Contre-indications for cytotoxic treatment according to the Summary of Product Characteristics (Arm B).
2. Clinical evidence of active brain metastasis or leptomeningeal involvement.
3. Other malignancy currently requiring active therapy.
4. QTc prolongation according to Fridericia formula deemed clinically relevant by the investigator (e.g., congenital long QT syndrome, QTc according to Fridericia formula > 470 ms).
5. Hypersensitivity to one of the trial drugs or the excipients.
6. Serious illness or concomitant non- oncological disease.
7. Systemic anticancer therapy within 4 weeks before the start of the study.
8. Evidence of ileus sor sub ileus.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (31):
- Belgium (4):
  - 1230.18.32003 Boehringer Ingelheim Investigational Site, Brussels
  - 1230.18.32004 Boehringer Ingelheim Investigational Site, Edegem
  - 1230.18.32002 Boehringer Ingelheim Investigational Site, Ghent
  - 1230.18.32001 Boehringer Ingelheim Investigational Site, Leuven
- France (15):
  - 1230.18.3321A Boehringer Ingelheim Investigational Site, Angers
  - 1230.18.3307A Boehringer Ingelheim Investigational Site, Bordeaux
  - 1230.18.3301A Boehringer Ingelheim Investigational Site, Caen
  - 1230.18.3322A Boehringer Ingelheim Investigational Site, Lille
  - 1230.18.3313A Boehringer Ingelheim Investigational Site, Lyon
  - 1230.18.3312A Boehringer Ingelheim Investigational Site, Nantes
  - 1230.18.3308A Boehringer Ingelheim Investigational Site, Nice
  - 1230.18.3302A Boehringer Ingelheim Investigational Site, Paris
  - 1230.18.3314A Boehringer Ingelheim Investigational Site, Paris
  - 1230.18.3309A Boehringer Ingelheim Investigational Site, Pierre-Bénite
  - 1230.18.3305A Boehringer Ingelheim Investigational Site, Reims
  - 1230.18.3320A Boehringer Ingelheim Investigational Site, Saint-Brieuc
  - 1230.18.3311A Boehringer Ingelheim Investigational Site, Strasbourg
  - 1230.18.3310A Boehringer Ingelheim Investigational Site, Toulouse
  - 1230.18.3315A Boehringer Ingelheim Investigational Site, Vandœuvre-lès-Nancy
- Slovakia (2):
  - 1230.18.42101 Boehringer Ingelheim Investigational Site, Bratislava
  - 1230.18.42103 Boehringer Ingelheim Investigational Site, Poprad
- Spain (7):
  - 1230.18.34006 Boehringer Ingelheim Investigational Site, Badalona
  - 1230.18.34001 Boehringer Ingelheim Investigational Site, Barcelona
  - 1230.18.34005 Boehringer Ingelheim Investigational Site, Barcelona
  - 1230.18.34007 Boehringer Ingelheim Investigational Site, Girona
  - 1230.18.34004 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1230.18.34002 Boehringer Ingelheim Investigational Site, Madrid
  - 1230.18.34003 Boehringer Ingelheim Investigational Site, Madrid
- Sweden (3):
  - 1230.18.46005 Boehringer Ingelheim Investigational Site, Linköping
  - 1230.18.46001 Boehringer Ingelheim Investigational Site, Stockholm
  - 1230.18.46003 Boehringer Ingelheim Investigational Site, Uppsala

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274
- [Derived] Pujade-Lauraine E, Selle F, Weber B, Ray-Coquard IL, Vergote I, Sufliarsky J, Del Campo JM, Lortholary A, Lesoin A, Follana P, Freyer G, Pardo B, Vidal L, Tholander B, Gladieff L, Sassi M, Garin-Chesa P, Nazabadioko S, Marzin K, Pilz K, Joly F. Volasertib Versus Chemotherapy in Platinum-Resistant or -Refractory Ovarian Cancer: A Randomized Phase II Groupe des Investigateurs Nationaux pour l'Etude des Cancers de l'Ovaire Study. J Clin Oncol. 2016 Mar 1;34(7):706-13. doi: 10.1200/JCO.2015.62.1474. Epub 2016 Jan 11. PMID 26755507

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall 54 patients were treated in Volasertib arm and 55 patients were treated in Cytotoxic arm. The "Not completed" category in the Subject Disposition table represents " Treatment permanently discontinued" and "The reasons for non-completion" in the table represent "Reason for treatment discontinuation".
Groups:
- Volasertib (BI 6727): Volasertib (BI 6727 300 mg) was administered as intravenous infusion over 2 hours at Day 1 of each 21-day treatment course.
  Treatment was to be administered until disease progression or occurrence of toxicity leading to treatment discontinuation. Patients withdrawn from volasertib treatment could receive a treatment according to investigator's choice. The patients were to be followed for survival status.
- Cytotoxic: Patients received a non-platinum cytotoxic single agent. The investigator chose the most appropriate drug according to patient status (previous chemotherapy effects, cumulative toxic effects, performance status, and nutritional status), the product Summary of Product Characteristics (SPC), and the local standard of care. The following non-platinum regimens were recommended because they are regarded efficacious and safe in patients with resistant ovarian cancer:
  * Pegylated liposomal doxorubicin (PLD): 40 mg/m² at Day 1 (1 course = 28 days)
  * Topotecan: 1.25 mg/m² from Days 1 to 5 (1 course = 21 days), or 4 mg/m² at Days 1, 8, and 15 (1 course = 28 days)
  * Paclitaxel: 80 mg/m² at Days 1, 8, 15, and 21 (1 course = 28 days)
  * Gemcitabine: 1000 mg/m² at Days 1 and 8 (1 course = 21 days)
Period: Overall Study
Arm/Group | Volasertib (BI 6727) | Cytotoxic
Started | 55 | 55 (24 patients switched to Volasertib (BI 6727) due to disease progression or occurrence of toxicity)
Completed | 0 | 0
Not Completed | 55 | 55
Not completed — Progressive disease RECIST | 44 | 28
Not completed — Wors. or AE of underlying cancer disease | 4 | 6
Not completed — Other AE | 3 | 10
Not completed — Non-compliant with protocol | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Refused continuation of study med. | 1 | 2
Not completed — Reason other than specified above | 2 | 6
Not completed — Not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set consisted of all patients who received at least one administration of the trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Volasertib (BI 6727) | Cytotoxic | Total
Number analyzed (Participants) | 54 | 55 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.88) | 60.9 (9.26) | 61.1 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 55 | 109
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR) at Week 24 According to Response Evaluation Criteria In Solid Tumours (RECIST) Version 1.1
Description: DCR was defined as the proportion of patients who had an overall response of complete response (CR), partial response (PR), or stable disease (SD).
Time Frame: Week 24
Population: TS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Volasertib (BI 6727) | Cytotoxic
Number analyzed (Participants) | 54 | 55
percentage of participants | 30.6 [18.0 to 43.2] | 43.1 [29.5 to 56.7]
Statistical Analysis 1: Comparison: Volasertib (BI 6727) vs Cytotoxic; Kaplan Meier estimates and confidence intervals (CI) were calculated using Greenwood's variance estimate within each treatment arm and the asymptotic CI for the difference in the rates found. The time was censored in those cases where there was no death or progression until the last trial visit; Test type: Superiority or Other; Difference in Kaplan-Meier DC rates = -12.5, 95% CI 2-sided [-31.1 to 6.0] — 95% CI using Greenwood´s variance estimate. Volasertib (BI 6727) minus Cytotoxic

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival of a patient was based on the investigator's assessment; it was defined as the number of days from the date of randomisation until the date of either disease progression or death from any cause, whichever occurred first.
  Definition of disease progression according to RECIST version 1.1; Patients with measurable tumour lesions at baseline, Target-lesions: at least a 20% increase in the sum of diameters of target lesions, the sum of diameters must also demonstrate an absolute increase of at least 5 mm,taking as reference the smallest sum on study, or appearance of 1 or more new lesions.
  Non-target lesions: unequivocal progression of existing non-target lesions or appearance of 1 or more new lesions Patients with non-measurable tumour lesions at baseline, Non-target lesions: requires unequivocal progression of existing non-target lesions or appearance of 1 or more new lesions
Time Frame: From randomization until disease progression, death or study discontinuation; Up to 213 weeks
Population: TS
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Volasertib (BI 6727) | Cytotoxic
Number analyzed (Participants) | 54 | 55
weeks | 13.1 [6.6 to 30.1] | 20.6 [11.6 to 30.7]
Statistical Analysis 1: Comparison: Volasertib (BI 6727) vs Cytotoxic; Test type: Superiority or Other; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.66 to 1.53] — Cox proportional-hazards regression model, stratified by disease status at baseline (measurable vs. non measurable disease) and platinum resistant vs platinum refractory disease at baseline. HR calculated as Volasertib (BI 6727) /Cytotoxic

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from randomisation to death irrespective of the cause of the death.
Time Frame: From randomization until death or study discontinuation; Up to 213 weeks
Population: TS
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Volasertib (BI 6727) | Cytotoxic
Number analyzed (Participants) | 54 | 55
weeks | 60.1 [31.3 to 95.4] | 68.6 [28.7 to 119.4]
Statistical Analysis 1: Comparison: Volasertib (BI 6727) vs Cytotoxic; Test type: Superiority or Other; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.63 to 1.42] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Best Overall Response
Description: Best overall response (BOR) is defined as the best response recorded at any time from the date of randomisation until the end of treatment.
  Missing categories signify that no tumour imaging has been performed post baseline, and therefore the response status could not be assessed.
Time Frame: time from the date of randomisation until study completion/discontinuation; Up to 213 weeks
Population: TS
Measure: Number; unit: participants
Arm/Group | Volasertib (BI 6727) | Cytotoxic
Number analyzed (Participants) | 54 | 55
participants
  CR- Measurable disease | 0 | 0
  PR- Measurable disease | 7 | 8
  SD- Measurable disease | 24 | 24
  PD- Measurable disease | 14 | 10
  Missing- Measurable disease | 0 | 2
  CR- Non-measurable disease | 0 | 1
  Non-CR/Non-PD- Non-measurable disease | 6 | 9
  PD- Non-measurable disease | 3 | 0
  Missing- Non-measurable disease | 0 | 1

5. Secondary Outcome: Biological Tumour Response Based on Serum Cancer Antigen 125 (CA-125) According to the Gynaecologic Cancer Intergroup (GCIG) Criteria
Description: Patients were to have a pre-treatment CA-125 of at least twice the upper limit of normal to be considered for CA-125 response. Patients were not evaluable by CA-125 if they had received mouse antibodies or if they had undergone medical and/or surgical interference with their peritoneum or pleura during the previous 28 days. In eligible patients, a CA-125 response was defined as the moment the CA- 25 was reduced by 50%, with this being confirmed with a consecutive CA-125 assessment not earlier than 28 days after the previous one.
  Biological response rate based on serum CA-125 levels was assessed according to the guidelines by the Gynaecologic Cancer Intergroup. Monitoring of blood levels of the tumour marker CA-125 was performed at screening and every 6 weeks thereafter.
Time Frame: At screening and every 6 weeks thereafter (Up to 213 weeks)
Population: TS
Measure: Number; unit: participants
Arm/Group | Volasertib (BI 6727) | Cytotoxic
Number analyzed (Participants) | 54 | 55
participants
  Yes | 10 | 12
  No | 33 | 23
  Not evaluable | 4 | 11
  Missing | 7 | 9

6. Secondary Outcome: Biological Progression-free Survival Based on Serum Cancer Antigen 125 (CA-125) According to the Gynaecologic Cancer Intergroup (GCIG) Criteria
Description: Biological PFS including assessment of CA-125 levels was defined as the time from randomisation until the first occurrence of progressive disease according to CA-125, progressive disease according to radiological evidence, or death.
  Also according to the below criterias,
  * In patients with radiological measurable disease, disease progression during study treatment could not be declared on the basis of CA-125 alone.
  * Patients with elevated CA-125 pre-treatment and normalization of CA-125 had to show evidence of CA-125 ≥ to two times the upper normal limit on two occasions at least one week apart or
  * Patients with elevated CA-125 pre-treatment, which never normalized, had to show evidence of CA-125 ≥ to two times the nadir value on two occasions at least one week apart or
  * Patients with CA-125 in the normal range pre-treatment had to show evidence of CA-125 ≥ to two times the upper normal limit on two occasions at least one week apart.
Time Frame: At screening and every 6 weeks thereafter (Up to 213 weeks )
Population: TS
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Volasertib (BI 6727) | Cytotoxic
Number analyzed (Participants) | 54 | 55
weeks | 13.1 [6.6 to 25.6] | 20.6 [11.6 to 30.0]
Statistical Analysis 1: Comparison: Volasertib (BI 6727) vs Cytotoxic; Test type: Superiority or Other; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.73 to 1.70] — Cox proportional-hazards regression model, stratified by disease status at baseline (measurable vs. non measurable disease) and platinum resistant vs platinum refractory disease at baseline. HR calculated as Volasertib (BI 6727)/ Cytotoxic

7. Secondary Outcome: Time to Deterioration in Global Health Status/Quality of Life (QOL)
Description: Time to deterioration in global health status/Quality of life (QOL) and symptom control assessed by the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30, QLQ-OV28, and individual symptom questionnaires.
  The time to deterioration was defined as the time from randomisation to a score increased (i.e. worsened) by at least 10 points from baseline (0-100 point scale). If score is missing, and patient died within 28 days after scheduled time for completion, the patient was considered deteriorated. In this case, time to deterioration is time to death.
Time Frame: Every 6 weeks (Up to 213 weeks )
Population: TS
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Volasertib (BI 6727) | Cytotoxic
Number analyzed (Participants) | 54 | 55
weeks | NA [12.3 to NA] — Missing median or percentiles signify that a sufficient number of events have not yet occurred to produce these estimates. | 39.6 [13.1 to 47.2]
Statistical Analysis 1: Comparison: Volasertib (BI 6727) vs Cytotoxic; Test type: Superiority or Other; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.40 to 1.61] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Time to Deterioration in Fatigue/Quality of Life (QOL)
Description: Time to deterioration in fatigue/Quality of life (QOL) and symptom control assessed by the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30, QLQ-OV28, and individual symptom questionnaires.
  The time to deterioration was defined as the time from randomisation to a score increased (i.e. worsened) by at least 10 points from baseline (0-100 point scale). If score is missing, and patient died within 28 days after scheduled time for completion, the patient was considered deteriorated. In this case, time to deterioration is time to death.
Time Frame: Every 6 weeks (Up to 213 weeks )
Population: TS
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Volasertib (BI 6727) | Cytotoxic
Number analyzed (Participants) | 54 | 55
weeks | NA [18.3 to NA] — Missing median or percentiles signify that a sufficient number of events have not yet occurred to produce these estimates. | 67.1 [12.4 to NA] — Missing median or percentiles signify that a sufficient number of events have not yet occurred to produce these estimates.
Statistical Analysis 1: Comparison: Volasertib (BI 6727) vs Cytotoxic; Test type: Superiority or Other; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.37 to 1.65] — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: Time to Deterioration in Pain/ Quality of Life (QOL)
Description: Time to deterioration in pain/ Quality of life (QOL) and symptom control assessed by the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30, QLQ-OV28, and individual symptom questionnaires.
  The time to deterioration was defined as the time from randomisation to a score increased (i.e. worsened) by at least 10 points from baseline (0-100 point scale). If score is missing, and patient died within 28 days after scheduled time for completion, the patient was considered deteriorated. In this case, time to deterioration is time to death.
Time Frame: Every 6 weeks (Up to 213 weeks )
Population: TS
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Volasertib (BI 6727) | Cytotoxic
Number analyzed (Participants) | 54 | 55
weeks | NA [16.6 to NA] — Missing median or percentiles signify that a sufficient number of events have not yet occurred to produce these estimates. | 54.1 [25.0 to NA] — Missing median or percentiles signify that a sufficient number of events have not yet occurred to produce these estimates.
Statistical Analysis 1: Comparison: Volasertib (BI 6727) vs Cytotoxic; Test type: Superiority or Other; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.39 to 1.93] — [estimate comment as in outcome 6, analysis 1]

10. Secondary Outcome: Time to Deterioration in Abdominal Bloating/ Quality of Life (QOL)
Description: Time to deterioration in abdominal bloating/ Quality of life (QOL) and symptom control assessed by the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30, QLQ-OV28, and individual symptom questionnaires.
  The time to deterioration was defined as the time from randomisation to a score increased (i.e. worsened) by at least 10 points from baseline (0-100 point scale). If score is missing, and patient died within 28 days after scheduled time for completion, the patient was considered deteriorated. In this case, time to deterioration is time to death.
Time Frame: Every 6 weeks (Up to 213 weeks )
Population: TS
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Volasertib (BI 6727) | Cytotoxic
Number analyzed (Participants) | 54 | 55
weeks | NA [12.9 to NA] — Missing median or percentiles signify that a sufficient number of events have not yet occurred to produce these estimates. | 47.2 [17.3 to 67.1]
Statistical Analysis 1: Comparison: Volasertib (BI 6727) vs Cytotoxic; Test type: Superiority or Other; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.33 to 1.47] — [estimate comment as in outcome 6, analysis 1]

11. Secondary Outcome: Time to Deterioration in the Three Most Troublesome Disease Specific Symptoms/ Quality of Life (QOL)
Description: Three most troublesome disease specific symptoms, defined by the patient at baseline.
  Patients that have defined more than 3 most troublesome symptoms have not been taken into account in the analysis.
  Quality of life (QOL) and symptom control assessed by the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30, QLQ-OV28, and individual symptom questionnaires.
  The time to deterioration was defined as the time from randomisation to a score increased (i.e. worsened) by at least 10 points from baseline (0-100 point scale). If score is missing, and patient died within 28 days after scheduled time for completion, the patient was considered deteriorated. In this case, time to deterioration is time to death.
Time Frame: Every 6 weeks (Up to 213 weeks)
Population: TS
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Volasertib (BI 6727) | Cytotoxic
Number analyzed (Participants) | 54 | 55
weeks | NA [NA to NA] — Missing median or percentiles signify that a sufficient number of events have not yet occurred to produce these estimates. | 18.9 [6.3 to NA] — Missing median or percentiles signify that a sufficient number of events have not yet occurred to produce these estimates.
Statistical Analysis 1: Comparison: Volasertib (BI 6727) vs Cytotoxic; Test type: Superiority or Other; Hazard Ratio (HR) = 0.27, 95% CI 2-sided [0.09 to 0.77] — [estimate comment as in outcome 6, analysis 1]

12. Secondary Outcome: Incidence and Intensity of Adverse Events According to the United States National Cancer Institute (US NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Description: Incidence and intensity of adverse events according to the United States National Cancer Institute (US NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0
Time Frame: From first treatment administration to 21 days after the last drug administration (Up to 1403 days)
Population: TS
Measure: Number; unit: participants
Groups:
- Cytotoxic to Volasertib Switch: Patients of the cytotoxic arm who switched to treatment with Volasertib (BI 6727).
Arm/Group | Volasertib (BI 6727) | Cytotoxic | Cytotoxic to Volasertib Switch
Number analyzed (Participants) | 54 | 55 | 24
participants
  Grade 1 | 4 | 3 | 1
  Grade 2 | 6 | 19 | 3
  Grade 3 | 16 | 25 | 9
  Grade 4 | 25 | 5 | 6
  Grade 5 | 3 | 3 | 3

13. Secondary Outcome: Clinically Relevant Changes in Laboratory and ECG Data
Description: Clinically relevant changes in laboratory and ECG data
Time Frame: From first treatment administration to 21 days after the last drug administration (Up to 1403 days)
Population: TS
Measure: Number; unit: percentage of participants
Arm/Group | Volasertib (BI 6727) | Cytotoxic | Cytotoxic to Volasertib Switch
Number analyzed (Participants) | 54 | 55 | 24
percentage of participants
  Blood alkaline phosphatase increased | 3.7 | 12.7 | 8.3
  Blood creatinine increased | 9.3 | 3.6 | 0.0
  Platelet count decreased | 9.3 | 0.0 | 8.3
  Alanine aminotransferase increased | 1.9 | 9.1 | 4.2
  Aspartate aminotransferase increased | 3.7 | 5.5 | 4.2
  Blood uric acid increased | 1.9 | 5.5 | 0.0
  Gamma-glutamyltransferase increased | 3.7 | 5.5 | 4.2
  Alanine aminotransferase abnormal | 0.0 | 0.0 | 4.2
  Electrocardiogram QT prolonged | 0.0 | 0.0 | 4.2
  Haemoglobin decreased | 3.7 | 3.6 | 4.2
  Neutrophil count decreased | 1.9 | 0.0 | 4.2
  Troponin I increased | 0.0 | 0.0 | 4.2
  Blood lactate dehydrogenase increased | 3.7 | 0.0 | 0.0
  Blood magnesium decreased | 3.7 | 0.0 | 0.0
  White blood cell count decreased | 3.7 | 0.0 | 0.0
  Blood urea increased | 1.9 | 3.6 | 0.0
  Alanine aminotransferase decreased | 1.9 | 0.0 | 0.0
  Blood bilirubin increased | 1.9 | 0.0 | 0.0
  Blood creatine phosphokinase decreased | 1.9 | 0.0 | 0.0
  Blood potassium decreased | 1.9 | 0.0 | 0.0
  Hepatic enzyme increased | 1.9 | 0.0 | 0.0
  Aspartate aminotransferase abnormal | 0.0 | 1.8 | 0.0
  Transaminases increased | 0.0 | 1.8 | 0.0

14. Secondary Outcome: AUC (0-24); Area Under the Concentration-time Curve in Plasma Over the Time Interval From 0 to 24 Hours for BI 6727 BS
Description: AUC (0-24); area under the concentration-time curve in plasma over the time interval from 0 to 24 hours for BI 6727 BS
Time Frame: -0.083 hours (h), 2h, 4h, 6h, 24h, 168h and 336 h after first drug administration
Population: All evaluable patients were to be included in the pharmacokinetic analysis. A patient was considered not evaluable if they had an important protocol violation relevant to the evaluation of pharmacokinetics or had insufficient data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Volasertib: Volasertib (BI 6727 300 mg) was administered as intravenous infusion over 2 hours at Day 1 of each 21-day treatment course.
  Treatment was to be administered until disease progression or occurrence of toxicity leading to treatment discontinuation. Patients withdrawn from volasertib treatment could receive a treatment according to investigator's choice. The patients were to be followed for survival status.
Arm/Group | Volasertib
Number analyzed (Participants) | 51
ng*h/mL | 2140 (25.5)

15. Secondary Outcome: AUC (0-24); Area Under the Concentration-time Curve in Plasma Over the Time Interval From 0 to 24 Hours for CD 10899 BS
Description: AUC (0-24); area under the concentration-time curve in plasma over the time interval from 0 to 24 hours for CD 10899 BS (metabolite of Volasertib BI 6727)
Time Frame: -0.083 hours (h), 2h, 4h, 6h, 24h, 168h and 336 h after first drug administration
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Volasertib
Number analyzed (Participants) | 51
ng*h/mL | 204 (65.3)

16. Secondary Outcome: AUC (0-inf); Area Under the Concentration-time Curve in Plasma Over the Time Interval From 0 Extrapolated to Infinity for BI 6727 BS
Description: AUC (0-inf); area under the concentration-time curve in plasma over the time interval from 0 extrapolated to infinity for BI 6727 BS
Time Frame: -0.083 hours (h), 2h, 4h, 6h, 24h, 168h and 336 h after first drug administration
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Volasertib
Number analyzed (Participants) | 49
ng*h/mL | 6240 (29.8)

17. Secondary Outcome: AUC (0-inf); Area Under the Concentration-time Curve in Plasma Over the Time Interval From 0 Extrapolated to Infinity for CD 10899 BS
Description: AUC (0-inf); area under the concentration-time curve in plasma over the time interval from 0 extrapolated to infinity for CD 10899 BS (metabolite of Volasertib BI 6727)
Time Frame: -0.083 hours (h), 2h, 4h, 6h, 24h, 168h and 336 h after first drug administration
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Volasertib
Number analyzed (Participants) | 51
ng*h/mL | 1400 (35.8)

18. Secondary Outcome: Cmax; Maximum Measured Concentration of BI 6727 BS in Plasma
Description: Cmax; maximum measured concentration of BI 6727 BS in plasma
Time Frame: -0.083 hours (h), 2h, 4h, 6h, 24h, 168h and 336 h after first drug administration
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Volasertib
Number analyzed (Participants) | 51
ng/mL | 341 (42.2)

19. Secondary Outcome: Cmax; Maximum Measured Concentration of CD 10899 BS in Plasma
Description: Cmax; maximum measured concentration of CD 10899 BS (metabolite of Volasertib BI 6727) in plasma
Time Frame: -0.083 hours (h), 2h, 4h, 6h, 24h, 168h and 336 h after first drug administration
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Volasertib
Number analyzed (Participants) | 51
ng/mL | 10.8 (63.4)

20. Secondary Outcome: Tmax; Time From Dosing to Maximum Measured Concentration of BI 6727 BS in Plasma
Description: tmax; time from dosing to maximum measured concentration of BI 6727 BS in plasma
Time Frame: -0.083 hours (h), 2h, 4h, 6h, 24h, 168h and 336 h after first drug administration
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | Volasertib
Number analyzed (Participants) | 51
hours | 2.00 [1.83 to 3.00]

21. Secondary Outcome: Tmax; Time From Dosing to Maximum Measured Concentration of CD 10899 BS in Plasma
Description: tmax; time from dosing to maximum measured concentration of CD 10899 BS (metabolite of Volasertib BI 6727) in plasma
Time Frame: -0.083 hours (h), 2h, 4h, 6h, 24h, 168h and 336 h after first drug administration
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | Volasertib
Number analyzed (Participants) | 51
hours | 6.07 [3.83 to 24.3]

22. Secondary Outcome: t1/2; Terminal Half-life of BI 6727 BS in Plasma
Description: t1/2; Terminal half-life of BI 6727 BS in plasma
Time Frame: -0.083 hours (h), 2h, 4h, 6h, 24h, 168h and 336 h after first drug administration
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Volasertib
Number analyzed (Participants) | 51
hours | 143 (21.3)

23. Secondary Outcome: t1/2; Terminal Half-life of CD 10899 BS in Plasma
Description: t1/2; Terminal half-life of CD 10899 BS in plasma
Time Frame: -0.083 hours (h), 2h, 4h, 6h, 24h, 168h and 336 h after first drug administration
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Volasertib
Number analyzed (Participants) | 53
hours | 146 (21.5)

24. Secondary Outcome: MRT; Mean Residence Time of BI 6727 BS in the Body
Description: MRT; Mean residence time of BI 6727 BS in the body
Time Frame: -0.083 hours (h), 2h, 4h, 6h, 24h, 168h and 336 h after first drug administration
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Volasertib
Number analyzed (Participants) | 49
hours | 118 (31.2)

25. Secondary Outcome: CL; Total Clearance of BI 6727 BS in Plasma After Intravenous Administration
Description: CL; total clearance of BI 6727 BS in plasma after intravenous administration
Time Frame: -0.083 hours (h), 2h, 4h, 6h, 24h, 168h and 336 h after first drug administration
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Volasertib
Number analyzed (Participants) | 49
mL/min | 801 (29.8)

26. Secondary Outcome: Vss;Apparent Volume of Distribution at Steady State Following Intravenous Administration for BI 6727 BS
Description: Vss;apparent volume of distribution at steady state following intravenous administration for BI 6727 BS
Time Frame: -0.083 hours (h), 2h, 4h, 6h, 24h, 168h and 336 h after first drug administration
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres
Arm/Group | Volasertib
Number analyzed (Participants) | 49
Litres | 5690 (25.8)

27. Secondary Outcome: Biomarkers and Pharmacogenetics Analysis (Optional)
Description: This endpoint has not been statistically analysed in the study report
Time Frame: 6 months
Arm/Group | Volasertib (BI 6727) | Cytotoxic
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first treatment administration to 21 days after the last drug administration (Up to 1403 days)
Arm/Group | Volasertib (BI 6727) | Cytotoxic | Cytotoxic to Volasertib Switch
Serious Adverse Events (participants affected / at risk) | 24/54 | 19/55 | 12/24
Other Adverse Events (participants affected / at risk) | 53/54 | 53/55 | 21/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib (BI 6727) (N=54) | Cytotoxic (N=55) | Cytotoxic to Volasertib Switch (N=24)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 2 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 3 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 0
Chest pain (General disorders) | 1 | 0 | 0
Condition aggravated (General disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0
Euthanasia (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Obstruction (General disorders) | 2 | 1 | 0
Pyrexia (General disorders) | 2 | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to heart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Panic reaction (Psychiatric disorders) | 1 | 0 | 0
Pyelocaliectasis (Renal and urinary disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Poor venous access (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib (BI 6727) (N=54) | Cytotoxic (N=55) | Cytotoxic to Volasertib Switch (N=24)
Anaemia (Blood and lymphatic system disorders) | 29 | 20 | 5
Leukopenia (Blood and lymphatic system disorders) | 15 | 8 | 2
Lymphopenia (Blood and lymphatic system disorders) | 7 | 8 | 0
Neutropenia (Blood and lymphatic system disorders) | 34 | 17 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 26 | 4 | 4
Abdominal distension (Gastrointestinal disorders) | 3 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 13 | 20 | 5
Abdominal pain upper (Gastrointestinal disorders) | 6 | 7 | 3
Ascites (Gastrointestinal disorders) | 1 | 3 | 2
Constipation (Gastrointestinal disorders) | 16 | 13 | 5
Diarrhoea (Gastrointestinal disorders) | 15 | 12 | 2
Dyspepsia (Gastrointestinal disorders) | 6 | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 19 | 25 | 5
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 3 | 0
Vomiting (Gastrointestinal disorders) | 15 | 18 | 2
Asthenia (General disorders) | 18 | 26 | 4
Chest pain (General disorders) | 4 | 2 | 1
Fatigue (General disorders) | 4 | 12 | 4
Mucosal inflammation (General disorders) | 4 | 7 | 1
Oedema peripheral (General disorders) | 8 | 5 | 3
Pain (General disorders) | 2 | 4 | 1
Pyrexia (General disorders) | 5 | 4 | 4
Hypersensitivity (Immune system disorders) | 2 | 0 | 2
Nasopharyngitis (Infections and infestations) | 4 | 2 | 1
Rhinitis (Infections and infestations) | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 2 | 5 | 0
Alanine aminotransferase increased (Investigations) | 1 | 5 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 7 | 2
Blood creatinine increased (Investigations) | 4 | 2 | 0
Blood uric acid increased (Investigations) | 1 | 3 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 3 | 1
Platelet count decreased (Investigations) | 5 | 0 | 2
Weight decreased (Investigations) | 4 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 11 | 14 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 5 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 4 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 7 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3
Dysgeusia (Nervous system disorders) | 1 | 4 | 0
Headache (Nervous system disorders) | 8 | 4 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 8 | 0
Paraesthesia (Nervous system disorders) | 3 | 4 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 3 | 0
Anxiety (Psychiatric disorders) | 1 | 4 | 1
Depression (Psychiatric disorders) | 0 | 3 | 1
Insomnia (Psychiatric disorders) | 4 | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 12 | 4
Erythema (Skin and subcutaneous tissue disorders) | 1 | 4 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights